CLINICAL TRIAL: NCT03675282
Title: Quantitative Mapping of Substantia Nigra Iron in Parkinson's Disease and Controls
Brief Title: Quantitative Mapping of Substantia Nigra Iron in Parkinson's Disease (Stages I-IV, REM Sleep Behavior Disorder) and Controls
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1711018740; 1R01NS095562-01A1 (NIH)
Record Dates: First submitted 2018-09-05; First posted 2018-09-18 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease; REM Sleep Behavior Disorder; Healthy
Keywords: MRI; PET Scan
MeSH Terms: conditions — Parkinson Disease; REM Sleep Behavior Disorder | interventions — N-(3-iodoprop-2-enyl)-2-beta-carbomethoxy-3-(4-methylphenyl)nortropane; Magnetic Resonance Spectroscopy; ioflupane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Parkinson Disease - Stage 1 (Experimental): MRI Brain at Baseline and 24 Months PE2i PET Scan or DaT Scan at Baseline and 24 Months Office Visit at Baseline and 24 Months
  Interventions: Drug: (11C)PE2I; Drug: Ioflupane
- Parkinson Disease - Stage 2 (Experimental): MRI Brain at Baseline and 24 Months PE2i PET Scan or DaT Scan at Baseline and 24 Months Office Visit at Baseline and 24 Months
  Interventions: Drug: (11C)PE2I; Drug: Ioflupane
- Parkinson Disease - Stage 3 (Experimental): MRI Brain at Baseline and 24 Months PE2i PET Scan or DaT Scan at Baseline and 24 Months Office Visit at Baseline and 24 Months
  Interventions: Drug: (11C)PE2I; Drug: Ioflupane
- Parkinson Disease - Stage 4 (Experimental): MRI Brain at Baseline and 24 Months PE2i PET Scan or DaT Scan at Baseline and 24 Months Office Visit at Baseline and 24 Months
  Interventions: Drug: (11C)PE2I; Drug: Ioflupane
- REM Sleep Behavior Disorder (Experimental): MRI Brain at Baseline and 24 Months PE2i PET Scan or DaT Scan at Baseline and 24 Months Office Visit at Baseline and 24 Months
  Interventions: Drug: (11C)PE2I; Drug: Ioflupane
- Healthy Controls (Experimental): MRI Brain at Baseline and 24 Months PE2i PET Scan or DaT Scan at Baseline and 24 Months Office Visit at Baseline and 24 Months
  Interventions: Drug: (11C)PE2I; Drug: Ioflupane

INTERVENTIONS:
Drug: (11C)PE2I — Subjects will received (11C)PE2I PET Scans at Baseline and 24 Month Visits
  Other Names: PET Scan
Drug: Ioflupane — Subjects will receive a DaT scan at baseline and 24 month visits if they don't receive a PE2I PET scan at baseline and 24 month visits
  Other Names: DaT scan

SUMMARY:
Prospective, single center study to determine whether the current R2* iron mapping method for measuring nigral iron changes in the brain can be significantly improved by using the Quantitative Susceptibility Mapping (QSM) based iron mapping techniques with the goal of validating QSM for potential use in later clinical trials. Subjects with a diagnosis of Parkinson's Disease, Rapid Eye Movement (REM) Sleep Behavior Disorder, and Normal Volunteers who meet the inclusion and exclusion criteria will be eligible for participation in this study.

DETAILED DESCRIPTION:
This study will evaluate the rate of iron accumulation throughout different stages of the disease and compare it to controls Thus, the investigators will be able to see if iron starts to accumulate in those patients, way before motor symptoms of Parkinson disease develop. Hypothetically, an iron chelator drug could remove excessive iron from the brain and slow down process of neurodegeneration. A precise technique to measure iron in the brain and to detect small changes therefore is needed as a radiological marker of disease progression and/or therapeutic effect in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* 1. Idiopathic Parkinson's Disease, REM Sleep Behavior Disorder subjects without signs of Parkinsonism and normal healthy controls a. If tremor is not present, subjects must have unilateral onset and persistent asymmetry of the symptoms. b. For PD Subjects only: Age > 30 years at time of diagnosis of PD with a maximum age of 100 years old c. Hoehn & Yahr stage < V (if PD)
* 2. For PD subjects only: Receiving an optimized dopaminergic regimen (i.e., either MAO-B inhibitor, a dopamine agonist and/or low doses of L-dopa, with dose change no more frequent than every 6-month in the course of the study); or medications naive
* 3. No overt anemia, iron deficiency, or other hematological disorders
* 4. Deemed healthy and able to undergo MRI and PE2i PET imaging by the Site Investigator, based on screening assessments-- medical history, physical examination 5. For Controls & REM Sleep Behavior Disorder Subjects Only: Age 20-80; willing to undergo multiple imaging sessions 6. Signed informed consent form

Exclusion Criteria:

* 1. Patient with atypical parkinsonism (such as suspected Progressive Supranuclear Palsy, Multiple System Atrophy) and secondary parkinsonism (such as normal pressure hydrocephalus, drug-induced, or vascular parkinsonism)
* 2. Patients with uncertainty as to having classical Parkinson's disease, such as those who might have scans without evidence of dopaminergic deficits (SWEDDs)
* 3. Presence of a medical or psychiatric comorbidity that can compromise participation in the study
* 4. Patients with clinically significant depression as determined by the Beck depression score > 15
* 5. History of exposure to typical or atypical neuroleptics or any dopamine blocking agent within 6 months prior to enrollment
* 6. Patients with psychosis/active hallucinations and memory difficulty pre-dating the onset of motor symptoms
* 7. History of brain surgery for PD
* 8. History of thyroid disease
* 9. History of stroke or cerebral vascular disease
* 10. History of drug abuse
* 11. History of repeated head injury or encephalitis
* 12. Positive dementia by DSM IV-R
* 13. Women of childbearing potential who are not surgically sterilized have to use a reliable measure of contraception and have a negative urine pregnancy test at the screening
* 14. Participation in other investigational drug trials within 30 days prior to screening
* 15. Contraindication for receiving MRI imaging such as presence of pacemakers, certain types of metallic implants, severe claustrophobia, history of reaction to contrast material, or renal insufficiency

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Shtilbans, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Parkinson Disease - Stage 1 | Parkinson Disease - Stage 2 | Parkinson Disease - Stage 3 | Parkinson Disease - Stage 4 | REM Sleep Behavior Disorder | Healthy Controls
Started | 20 | 27 | 2 | 0 | 9 | 24
Completed | 15 | 17 | 1 | 0 | 7 | 17
Not Completed | 5 | 10 | 1 | 0 | 2 | 7
Not completed — Lost to Follow-up | 4 | 8 | 1 | 0 | 2 | 7
Not completed — received clinical care that was exclusionary to the study | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 0 subjects were analyzed in the PD Stage 4 arm because no Stage 4 patients were enrolled
Groups:
- Total: Total of all reporting groups
Arm/Group | Parkinson Disease - Stage 1 | Parkinson Disease - Stage 2 | Parkinson Disease - Stage 3 | Parkinson Disease - Stage 4 | REM Sleep Behavior Disorder | Healthy Controls | Total
Number analyzed (Participants) | 20 | 27 | 2 | 0 | 9 | 24 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (7.9) | 67.7 (8.8) | 75.0 (2.8) |  | 59.6 (2.9) | 61.5 (8.6) | 64.2 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 0 |  | 1 | 9 | 24
  Male | 14 | 19 | 2 |  | 8 | 15 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 |  | 2 | 1 | 4
  Not Hispanic or Latino | 13 | 16 | 2 |  | 5 | 15 | 51
  Unknown or Not Reported | 6 | 11 | 0 |  | 2 | 8 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 |  | 0 | 0 | 0
  Asian | 0 | 0 | 0 |  | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 |  | 0 | 6 | 6
  White | 11 | 16 | 2 |  | 7 | 5 | 41
  More than one race | 0 | 0 | 0 |  | 0 | 0 | 0
  Unknown or Not Reported | 9 | 11 | 0 |  | 2 | 12 | 34
MOCA score [Mean (Standard Deviation); unit: scores on a scale] — The Montreal Cognitive Assessment (MOCA) is a brief test that screens for cognitive impairment and dementia. The lowest score is 0 and the highest score is 30. A score of 26 or higher is generally considered normal, while lower scores indicate cognitive impairment.
  scores on a scale | 26.5 (2.1) | 25.6 (3.6) | 29 (0) |  | 27.4 (1.7) | 26.3 (1.9) | 26.3 (2.6)
UPDRS Scores [Mean (Standard Deviation); unit: scores on a scale] — The Unified Parkinson's Disease Rating Scale (UPDRS) is a tool used to measure the severity and progression of Parkinson's disease.
  Part I: evaluation of mentation, behavior, and mood (0-16) Part II: self-evaluation of the activities of daily life (ADLs) including speech, swallowing, handwriting, dressing, hygiene, falling, salivating, turning in bed, walking, and cutting food (0-52) Part III: clinician-scored monitored motor evaluation (0-108) Part IV: complications of therapy (0-23)
  The higher the score value, the worse symptoms are.
  scores on a scale
    UPDRS Part I | 2.25 (1.83) | 1.88 (1.67) | 5 (0.0) |  | 1.67 (1.50) | 0.91 (2.57) | 1.71 (2.06)
    UPDRS Part II | 6.11 (4.42) | 7.28 (4.63) | 13 (0) |  | 0.56 (1.01) | 0 (0) | 4.10 (4.84)
    UPDRS Part III | 16.6 (6.3) | 24.0 (10.3) | 34 (0) |  | 0.6 (1.1) | 0 (0) | 12.4 (12.7)
    UPDRS Part IV | 2.63 (1.89) | 2.80 (3.33) | 0 (0) |  | 0.78 (0.83) | 0.09 (0.29) | 1.68 (2.45)
Sensitivity of QSM MR Imaging [Mean (Standard Deviation); unit: ppb] | 379.5896 (84.4375) | 314.1832 (138.1896) | 561.1894 (0.0) |  | 288.1832 (122.8809) | 261.6498 (72.7075) | 314.6444 (117.1813)
PE2i PET scan [Mean (Standard Deviation); unit: Bmax/Kd] | 3.47 (1.30) | 3.10 (1.20) | 2.33 (0.0) |  | 3.87 (0.95) | 3.58 (1.37) | 3.39 (1.25)

OUTCOME MEASURES:

1. Primary Outcome: Change in Sensitivity of QSM MR Imaging From Baseline MR Imaging to 24 Month MR Imaging
Description: Change in Sensitivity of QSM MR imaging as compared to R2* from baseline MR imaging to 24 month MR imaging, as measured by Radiology reader agreements
Time Frame: Baseline and 24 Months
Population: This analysis population included Parkinson's disease patients, stages I-III, REM Sleep behavior disorder patients, and healthy controls who completed the study. One Stage III Parkinson's disease patient was excluded because their MRI protocol did not include T1, and we were therefore unable to get QSM values. 0 subjects were analyzed for the PD Stage 4 arm because no Stage 4 patients were enrolled.
Measure: Mean (Standard Deviation); unit: ppb
Arm/Group | Parkinson Disease - Stage 1 | Parkinson Disease - Stage 2 | Parkinson Disease - Stage 3 | Parkinson Disease - Stage 4 | REM Sleep Behavior Disorder | Healthy Controls
Number analyzed (Participants) | 15 | 17 | 1 | 0 | 7 | 17
ppb
  Baseline | 379.5896 (84.4375) | 314.1832 (138.1896) | 561.1894 (0) |  | 288.1832 (122.8809) | 261.6498 (72.7075)
  24 Months | 359.7905 (152.2746) | 335.4785 (117.6937) | 0.0 (0.0) |  | 287.3132 (141.0688) | 250.1543 (80.9845)
Statistical Analysis 1: Comparison: Parkinson Disease - Stage 1; Parkinson Disease - Stage 1 (Baseline vs. 24 months); Test type: Superiority; p = 0.66, paired t-test; Mean Difference (Final Values) = 19.8
Statistical Analysis 2: Comparison: Parkinson Disease - Stage 2; Parkinson Disease - Stage 2 (Baseline vs. 24 months); Test type: Superiority; p = 0.63, paired t-test; Mean Difference (Final Values) = -21.3
Statistical Analysis 3: Comparison: REM Sleep Behavior Disorder; REM Sleep Behavior Disorder (Baseline vs. 24 months); Test type: Superiority; p = 0.99, paired t-test; Mean Difference (Final Values) = 0.87
Statistical Analysis 4: Comparison: Healthy Controls; Healthy Controls (Baseline vs. 24 months); Test type: Superiority; p = 0.67, paired t-test; Mean Difference (Final Values) = 11.5

2. Secondary Outcome: Assess Clinical Changes in Disease Arm
Description: Assess clinical changes in disease arm, as measured by changes in unified Parkinson's disease rating scale (UPDRS) scale assessments at baseline and 24 Month visits. The UPDRS is used to follow the longitudinal course of Parkinson's disease.
  The UPDRS is made up of 42 questions grouped into 4 sections:
  Part I: evaluation of mentation, behavior, and mood Part II: self-evaluation of the activities of daily life (ADLs) including speech, swallowing, handwriting, dressing, hygiene, falling, salivating, turning in bed, walking, and cutting food Part III: clinician-scored monitored motor evaluation Part IV: complications of therapy
  score for part I range is: 0-16 score for part II range is:0- 52 score for part III range is: 0-108 score for part IV range is: 0-23
  The higher the score value, the worse symptoms are.
Time Frame: Baseline and 24 Months
Population: This analysis population included Parkinson's disease patients, stages I-III, REM Sleep behavior disorder patients, and healthy controls who completed the study. 0 subjects were analyzed for the PD Stage 4 arm because no Stage 4 patients were enrolled
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parkinson Disease - Stage 1 | Parkinson Disease - Stage 2 | Parkinson Disease - Stage 3 | Parkinson Disease - Stage 4 | REM Sleep Behavior Disorder | Healthy Controls
Number analyzed (Participants) | 15 | 17 | 1 | 0 | 7 | 17
score on a scale
  UPDRS Part I: Baseline | 2.25 (1.83) | 1.88 (1.67) | 5 (0) |  | 1.67 (1.50) | 0.91 (2.57)
  UPDRS Part II: Baseline | 6.11 (4.42) | 7.28 (4.63) | 13 (0) |  | 0.56 (1.01) | 0 (0)
  UPDRS Part III: Baseline | 16.6 (6.3) | 24.0 (10.3) | 34 (0) |  | 0.6 (1.1) | 0 (0)
  UPDRS Part IV: Baseline | 2.63 (1.89) | 2.80 (3.33) | 0 (0) |  | 0.78 (0.83) | 0.09 (0.29)
  UPDRS Part I: 24 Months | 2.875 (2.156) | 2.294 (2.144) | 11.0 (0.0) |  | 2.857 (1.464) | 0.706 (1.404)
  UPDRS Part II: 24 Months | 7.563 (4.899) | 9.059 (6.722) | 31.0 (0.0) |  | 0.714 (0.756) | 0.529 (0.80)
  UPDRS Part III: 24 Months | 22.75 (9.248) | 27.588 (6.643) | 42.0 (0.0) |  | 1.429 (1.618) | 0.0 (0.0)
  UPDRS Part IV: 24 Months | 2.686 (1.922) | 3.176 (2.834) | 3.0 (0.0) |  | 0.857 (0.690) | 0.471 (0.624)
Statistical Analysis 1: Comparison: Parkinson Disease - Stage 1; Parkinson Disease - Stage 1 UPDRS Part I (Baseline vs. 24 months); Test type: Superiority; p = 0.40, paired t-test; Mean Difference (Final Values) = -0.625
Statistical Analysis 2: Comparison: Parkinson Disease - Stage 1; Parkinson Disease - Stage 1 UPDRS Part II (Baseline vs. 24 months); Test type: Superiority; p = 0.40, paired t-test; Mean Difference (Final Values) = -1.453
Statistical Analysis 3: Comparison: Parkinson Disease - Stage 1; Test type: Superiority; p = 0.04, paired t-test — Parkinson Disease - Stage 1 UPDRS Part III (Baseline vs. 24 months); Mean Difference (Final Values) = -6.15
Statistical Analysis 4: Comparison: Parkinson Disease - Stage 1; Parkinson Disease - Stage 1 UPDRS Part IV (Baseline vs. 24 months); Test type: Superiority; p = 0.94, paired t-test; Mean Difference (Final Values) = -0.056
Statistical Analysis 5: Comparison: Parkinson Disease - Stage 2; Parkinson Disease - Stage 2 UPDRS Part I (Baseline vs. 24 months); Test type: Superiority; p = 0.53, paired t-test; Mean Difference (Final Values) = -0.414
Statistical Analysis 6: Comparison: Parkinson Disease - Stage 2; Parkinson Disease - Stage 2 UPDRS Part II (Baseline vs. 24 months); Test type: Superiority; p = 0.38, paired t-test; Mean Difference (Final Values) = -1.779
Statistical Analysis 7: Comparison: Parkinson Disease - Stage 2; Parkinson Disease - Stage 2 UPDRS Part III (Baseline vs. 24 months); Test type: Superiority; p = 0.24, paired t-test; Mean Difference (Final Values) = -3.59
Statistical Analysis 8: Comparison: Parkinson Disease - Stage 2; Parkinson Disease - Stage 2 UPDRS Part IV (Baseline vs. 24 months); Test type: Superiority; p = 0.73, paired t-test; Mean Difference (Final Values) = -0.376
Statistical Analysis 9: Comparison: REM Sleep Behavior Disorder; REM Sleep Behavior Disorder UPDRS Part I (Baseline vs. 24 months); Test type: Superiority; p = 0.16, paired t-test; Mean Difference (Final Values) = -1.187
Statistical Analysis 10: Comparison: REM Sleep Behavior Disorder; REM Sleep Behavior Disorder UPDRS Part II (Baseline vs. 24 months); Test type: Superiority; p = 0.75, paired t-test; Mean Difference (Final Values) = -0.154
Statistical Analysis 11: Comparison: REM Sleep Behavior Disorder; REM Sleep Behavior Disorder UPDRS Part III (Baseline vs. 24 months); Test type: Superiority; p = 0.28, paired t-test; Mean Difference (Final Values) = -0.829
Statistical Analysis 12: Comparison: REM Sleep Behavior Disorder; REM Sleep Behavior Disorder UPDRS Part IV (Baseline vs. 24 months); Test type: Superiority; p = 0.85, paired t-test; Mean Difference (Final Values) = -0.077
Statistical Analysis 13: Comparison: Healthy Controls; Healthy Controls UPDRS Part I (Baseline vs. 24 months); Test type: Superiority; p = 0.78, paired t-test; Mean Difference (Final Values) = 0.204
Statistical Analysis 14: Comparison: Healthy Controls; Healthy Controls UPDRS Part IV (Baseline vs. 24 months); Test type: Superiority; p = 0.03, paired t-test; Mean Difference (Final Values) = -0.381

3. Secondary Outcome: Assess Change in PE2i PET Scan or DaT Scan
Description: Assess changes in dopamine depletion as measured by the baseline PE2i PET scan or DaT scan compared to the 24 month PE2i PET scan or DaT scan
Time Frame: Baseline and 24 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Bmax/Kd
Arm/Group | Parkinson Disease - Stage 1 | Parkinson Disease - Stage 2 | Parkinson Disease - Stage 3 | Parkinson Disease - Stage 4 | REM Sleep Behavior Disorder | Healthy Controls
Number analyzed (Participants) | 15 | 17 | 1 | 0 | 7 | 17
Bmax/Kd
  Baseline | 3.47 (1.30) | 3.10 (1.20) | 2.33 (0.0) |  | 3.87 (0.95) | 3.58 (1.37)
  24 Months | 3.07 (0.65) | 3.07 (1.17) | 2.38 (0) |  | 3.37 (1.41) | 3.48 (0.80)
Statistical Analysis 1: Comparison: Parkinson Disease - Stage 1; Parkinson Disease - Stage 1 (Baseline vs. 24 months); Test type: Superiority; p = 0.30, paired t-test; Mean Difference (Final Values) = 0.40
Statistical Analysis 2: Comparison: Parkinson Disease - Stage 2; Parkinson Disease - Stage 2 (Baseline vs. 24 months); Test type: Superiority; p = 0.94, paired t-test; Mean Difference (Final Values) = 0.03
Statistical Analysis 3: Comparison: REM Sleep Behavior Disorder; REM Sleep Behavior Disorder (Baseline vs. 24 months); Test type: Superiority; p = 0.45, paired t-test; Mean Difference (Final Values) = 0.50
Statistical Analysis 4: Comparison: Healthy Controls; Healthy Controls (Baseline vs. 24 months); Test type: Superiority; p = 0.80, paired t-test; Mean Difference (Final Values) = 0.10

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the course of the study per participant which was 2 years ± 2 months.
Description: The number of participants in Parkinson's disease Stage 4 arm for serious adverse events, all cause mortality, and other adverse events are all zero because we did not recruit any PD stage 4 patients.
Groups:
- Parkinson's Disease Stage 1: PD stage 1
- Parkinson's Disease Stage 2: PD stage 2
- Parkinson's Disease Stage 3: PD stage 3
- Parkinson's Disease Stage 4: PD stage 4
- REM Sleep Behavior Disorder: RBD
- Healthy Controls: Healthy controls
Arm/Group | Parkinson's Disease Stage 1 | Parkinson's Disease Stage 2 | Parkinson's Disease Stage 3 | Parkinson's Disease Stage 4 | REM Sleep Behavior Disorder | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/27 | 0/2 | 0/0 | 0/9 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/27 | 0/2 | 0/0 | 0/9 | 0/24
Other Adverse Events (participants affected / at risk) | 0/20 | 0/27 | 0/2 | 0/0 | 0/9 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT03675282/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/82/NCT03675282/ICF_000.pdf